CLINICAL TRIAL: NCT05395520
Title: Vancomycin Monitoring: Is AUC Monitoring Appropriate for More Than Just Serious MRSA Infections?
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 007.PHA.2021.C
Record Dates: First submitted 2022-04-27; First posted 2022-05-27 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-07

CONDITIONS: MRSA

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Retrospective chart review — Retrospective chart review to be conducted at Methodist Charlton Medical Center (MCMC) in Dallas, TX. Adult patients who received vancomycin while inpatient at MCMC with at least one corresponding vancomycin trough level taken at steady state will be included. All vancomycin orders by providers are entered as pharmacy to dose; thus dosing and routine monitoring is conducted by pharmacists.

SUMMARY:
Vancomycin, a glycopeptide antibiotic, is commonly prescribed as initial therapy for hospitalized patients due to its broad gram-positive coverage. Vancomycin is used for the treatment and prevention of a variety of bacterial infections ranging from streptococcal to methicillin-resistant Staphylococcus aureus (MRSA) infections.1 Notable adverse effects of intravenous vancomycin include nephrotoxicity, ototoxicity and hypersensitivity reactions. Given its pharmacokinetic profile, therapeutic drug monitoring is essential in determining the therapeutic efficacy of vancomycin as well as for avoiding nephrotoxicity.

DETAILED DESCRIPTION:
Vancomycin, a glycopeptide antibiotic, is commonly prescribed as initial therapy for hospitalized patients due to its broad gram-positive coverage. Vancomycin is used for the treatment and prevention of a variety of bacterial infections ranging from streptococcal to methicillin-resistant Staphylococcus aureus (MRSA) infections.1 Notable adverse effects of intravenous vancomycin include nephrotoxicity, ototoxicity and hypersensitivity reactions. Given its pharmacokinetic profile, therapeutic drug monitoring is essential in determining the therapeutic efficacy of vancomycin as well as for avoiding nephrotoxicity.

The 2020 guidelines continue to enforce AUC/MIC as the preferred PK/PD parameter, but now recommend utilizing vancomycin peak and trough concentrations to target an AUC/MIC of 400-600 mg*h/L for serious MRSA infections. Although this AUC goal is not new, the 2009 consensus guidelines previously recommended trough only monitoring as a simplistic surrogate marker for attaining this AUC goal. Furthermore, the most accurate way of calculating AUC requires obtaining two steady state vancomycin serum concentrations over one dosing period. In this way, AUC guided monitoring requires more pharmacist and nursing time, the use of more hospital resources and additional cost to the patient.

As was true of the 2009 guidelines, the 2020 guidelines also leave certain questions unanswered. The paucity and conflicting data of vancomycin monitoring in patients with non-serious MRSA infections (skin and soft tissue infections, urinary tract infections, etc.), methicillin-sensitive Staphylococcus aureus (MSSA) infections and non-staphylococcal pathogen infections has left no guidance on the ideal vancomycin PK/PD targets in these patient populations. A literature search of AUC/MIC monitoring in patients with streptococcal and enterococcal infections yielded very few studies in patients with enterococcal infections and no studies in patients with streptococcal infections.

ELIGIBILITY:
Inclusion Criteria:

* Patients hospitalized from June 2020- January 2021.
* 18 years and older
* At least 1 vancomycin trough concentration drawn at steady state
* Organism with an MIC of 2 mg/L, if vancomycin was continued and in whom a steady state trough concentration was obtained

Exclusion Criteria:

* Patients with end stage renal disease (on hemodialysis or peritoneal dialysis) or on continuous renal replacement therapy

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients who received vancomycin while inpatient at MCMC with at least one corresponding vancomycin trough level taken at steady state will be included.
Sampling Method: Non-Probability Sample
Enrollment: 146 (Estimated)
Dates: Start 2021-04-08 (Actual); Primary Completion 2024-04-08 (Estimated); Study Completion 2024-04-08 (Estimated)

PRIMARY OUTCOMES:
Efficacy of trough and AUC vancomycin monitoring | up to 1 year
  To compare the efficacy of targeting troughs of 10-20 mg/L vs targeting AUC of 400-600 for vancomycin monitoring without the use of vancomycin peak serum concentrations. o AUC will be calculated via the trapezoidal method.o Troughs will be stratified in the following categories: < 10 mg/L, 10-15 mg/L, 15-20 mg/L and > 20 mg/L.
• Determine differences in efficacy/clinical outcome and re-admission rates of AUC monitoring compared to trough monitoring in severe or deep-seeded infections (pneumonia, endocarditis, osteomyelitis or bacteremia) | up to 1 year
  Readmission rate of AUC monitoring compared to trough monitoring. Re-admission within 30 days will be classified as due to previous infection or all-cause.

CONTACTS AND LOCATIONS:
Overall Officials: Akins Ronda, PharmD, Principal Investigator — Methodist Health System
Locations (1):
- Methodist Dallas Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No